CLINICAL TRIAL: NCT07050238
Title: SAFEGUARD Life Force
Brief Title: Evaluation of a Group-based, Skills Training for Increasing Mental Toughness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Defense Health Agency (U.S. Federal Agency); Harvard University (Other); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Regents of the University of Michigan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USUHS.2025-152
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: Resilience; Mental Toughness
Keywords: Mental Toughness; Active-duty Military; Risk Reduction; Prevention
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life Force program (Experimental): The Life Force program is a 5-session, group-based, skills training program tailored specifically for active duty Soldiers. The program uses evidence-based strategies to mitigate harmful and high-risk behaviors and promote Mental Toughness.
  Interventions: Behavioral: Life Force
- Control (No Intervention): Standard of care with 6- and 12-month follow up assessments.

INTERVENTIONS:
Behavioral: Life Force — 5-session, group-based, skills training program tailored specifically for active-duty Soldiers aimed at mitigating harmful and high-risk behaviors and promote Mental Toughness.
  Arms: Life Force program

SUMMARY:
The goal of the Life Force study is to (1) evaluate the efficacy of targeted, skills-based training for enhancing mental toughness and mitigating harmful and high-risk behaviors in active-duty Soldiers, and (2) to determine who benefits the most from this type of training. Researchers will compare the training group to a control group. All participants will complete a baseline survey and two follow up surveys at 6 and 12 months post-baseline. The group assigned to the Life Force training condition will also complete a 5-session, group-based, skills training program.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of the Life Force training program, a 5- session, group-based, skills training program tailored specifically for active-duty Soldiers. The program uses evidence-based strategies to mitigate harmful and high-risk behaviors and promote Mental Toughness-defined as the ability to maintain peak performance under pressure or adversity, recover from setbacks, cope effectively with challenges, maintain a positive attitude, and persevere towards goals. The training sessions are led by skilled Life Force trainers from the study team and focus on building the following skills:

* Grow Through Support - building the inner circle and recognizing when to lean on that support
* Relentlessness - mastering the ability to push forward past the point of quitting
* Invite Adversity - fail forward, seeing failure as an opportunity for growth
* Nonstop Resolve - owning the setback, taking accountability of mistakes to reset and move forward
* Dominate Your Emotions - controlling emotions, breaking down intervention points and how to respond instead of reacting Participants will complete a 15-20 minute baseline survey. An AI machine learning algorithm, built from existing military administrative and health records, will be used to determine eligibility for participation by predicting who will benefit most from this training. Eligible participants will be randomly assigned to either the Life Force training or a control group. The training group will participate in 5 group training sessions. Both the training and control groups will complete two 15-20 minute follow-up surveys at 6 and 12 months. The surveys will assess for the occurrence of high-risk behaviors or events qualified for an Army Serious Incident Report (SIR), indicators of poor performance, and self-reported improvements in mental toughness, military readiness, job satisfaction, career intentions, and overall functioning in their occupational, personal, and social lives. Training group data will be compared to the control group (who will only complete the surveys).

ELIGIBILITY:
Inclusion Criteria:

* Active duty Soldiers in the regular Army
* Age 18 or older
* Stationed at Fort Hood, TX

Exclusion Criteria:

* Soldiers with self-identified plans of leaving active duty service within 12 months of the baseline assessment
* Soldiers having a planned permanent change in station (PCS) or deployment within 12 months of the baseline assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Risky/Harmful Behaviors | Within the 12 months following completion of the baseline assessment
  Self-reported or administratively recorded

SECONDARY OUTCOMES:
Poor Performance | Within the 12 months following completion of the baseline assessment
  Poor performance as indicated either by written reprimands, designations in the NCOER, a corrective action plan (DA Form 4856), remedial training, flagging actions, demotion, Article 15, or barred reenlistment
Mental Toughness | Within the 12 months following completion of the baseline assessment
  Self-reported; From the Sports Mental Toughness Questionnaire
Military Readiness, Satisfaction, & Career Plans | Within the 12 months following completion of the baseline assessment
  Self-reported
Suicide-related behaviors | Within the 12 months following completion of the baseline assessment
  Self-reported
Role Functioning (occupational, personal, and social) | Within the 12 months following completion of the baseline assessment
  Self-reported

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Hood, Killeen, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided